CLINICAL TRIAL: NCT02531048
Title: Normative Values Laser Nociceptive Evoked Potentials Depending on the Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0701035; 2007- A00535-48 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-20; First posted 2015-08-21 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2016-03

CONDITIONS: Healthy
Keywords: healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteers (Experimental): Healthy volunteers are able to participate to this study. They must not have neurological troubles. They will have different stimulations :
  * laser stimulations on lower limbs
  * laser stimulations cervical
  * 20 laser stimulations for each site on the upper limbs
  * laser stimulations on face and neck
  Interventions: Device: laser stimulations on lower limbs; Device: laser stimulations cervical; Device: 20 laser stimulations for each site on the upper limbs; Device: laser stimulations on face and neck

INTERVENTIONS:
Device: laser stimulations on lower limbs — 20 laser stimulations for each site : back foot, outer face of the legs, and anterior thigh
Device: laser stimulations cervical — 15 laser stimulations cervical areas below the ears.
Device: 20 laser stimulations for each site on the upper limbs — 20 laser stimulations for each site : back of the hands and arms front face
Device: laser stimulations on face and neck — 15 lasers stimulations for each site : mandibular areas and areas below the ears.

SUMMARY:
Different neurological damage may alter the pain conduction systems centrally (spinothalamic pathway) or peripherally (small caliber sensory fibers A delta and C). The laser thermal stimulation selectively stimulates the pain pathways and generates nociceptive signals conveyed to the cortex. Registering these cortical responses constitute the technical laser nociceptive evoked potentials. If these tests are routinely used, their interpretation must remain cautious especially in the elderly.

DETAILED DESCRIPTION:
Different neurological damage may alter the pain conduction systems centrally (spinothalamic pathway) or peripherally (small caliber sensory fibers A delta and C). The laser thermal stimulation selectively stimulates the pain pathways and generates nociceptive signals conveyed to the cortex. Registering these cortical responses constitute the technical laser nociceptive evoked potentials. If these tests are routinely used, their interpretation must remain cautious especially in the elderly. Normal values that are available have been obtained in young subjects. However, various studies have shown that the integration of nociceptive messages depended on age. The aim of this study was to establish normal values of nociceptive evoked potentials for each age group of 18 to 75 years.

ELIGIBILITY:
Inclusion Criteria:

* major

Exclusion Criteria:

* Neurological history
* Neuralgia history (> 3 months)
* Pathology can cause neuropathy (unbalanced thyroid dysfunction, diabetes, kidney failure, chronic hepatitis, HIV ...)
* Dermatological disorder known type of Lucite or photosensitivity
* Medical treatment analgesic, psychotropic or anti-epileptic underway
* Toxic acquired in the last 72 hours (alcohol, cannabis, other toxic ...)
* Pregnant women
* Incapacitate to stand still
* Participation in another biomedical research in the field of pain in the three months prior to inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2012-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
composite outcomes : latencies (ms) and amplitudes (μV) of nociceptive evoked potential | Day 0

SECONDARY OUTCOMES:
detection threshold (mJ/mm2) | Day 0
nociceptive threshold (mJ/mm2) | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Creac'h, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No